CLINICAL TRIAL: NCT06135792
Title: The Effect of Arginine on Biofilm Composition, Architecture and Metabolism in Caries-active Patients: a Split-mouth in Situ Trial
Brief Title: The Effect of Arginine on Biofilm Composition, Architecture and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 97473
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries; Dental Plaque; Microbial Colonization
MeSH Terms: conditions — Dental Caries; Dental Plaque; Communicable Diseases | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arginine solution (Experimental): Arginine treatment is performed outside the oral cavity (ex vivo) by immersing one side of a splint into a solution of arginine 1.5% (w/v). Treatment is performed 3 times a day for 30 min.
  Interventions: Other: Arginine
- Placebo (Placebo Comparator): Placebo treatment is performed outside the oral cavity (ex vivo) by immersing one side of a splint into distilled water. Treatment is performed 3 times a day for 30 min.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Arginine — See arm description
  Arms: Arginine solution
Other: Placebo — See arm description
  Arms: Placebo

SUMMARY:
Arginine is an adjunct to oral health care that has the potential to modulate the composition and activity of the microbial community of dental biofilms towards a health-related status without harmful effects for the resident oral microbiota. The aim of the study is to investigate the effects of arginine treatment compared to placebo on the composition, metabolism, and microarchitecture of biofilms grown in situ in the oral cavity of caries-active participants.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years old.
* Three or more active carious lesions.
* Anatomically possible to manufacture an intraoral lower-jaw splint.
* Able to understand and follow instructions, as well as to read and sign the informed consent form.

Exclusion Criteria:

* History of allergies towards any of the ingredients in the test products
* Self-reported pregnant or nursing
* Antibiotic or anti-inflammatory medication within 90 days of the screening visit.
* Orthodontic appliances, including retainers, or removable partial dentures.
* Self-reported serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Biofilm pH | Measured after in situ biofilm growth
  Extracellular biofilm pH measured after sucrose challenge using pH ratiometry

SECONDARY OUTCOMES:
Biofilm microbial composition | Analyzed after in situ biofilm growth
  Microbial community of dental biofilms determined by 16S rRNA gene sequencing. Distribution of specific microbial targets in the biofilms is visualized by fluorescence in situ hybridization.
Biofilm matrix architecture | Analyzed after of in situ biofilm growth
  Matrix components are visualized in the dental biofilms by confocal microscopy.
Biofilm thickness | Measured after in situ biofilm growth
  Measured using confocal laser scanning microscopy and/or optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schlafer, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to general data protection regulations, individual participant data will not be made available publicly. Summary data will be made available upon publication of the results.